CLINICAL TRIAL: NCT04442139
Title: Patient Reported Outcomes of a "Tailored" Bilio-Pancreatic Limb Length on Mean Weight Loss and Mean Daily Dietary Food Choices in the One Anastomosis Gastric Bypass (Mini-Gastric Bypass-Original Technique)
Brief Title: Patient Reported Outcomes of a "Tailored" Bilio-Pancreatic Limb Length on Daily Food Choices in Mini-Gastric Bypass
Acronym: TaBLFood-MGB
Status: Completed | Type: Observational
Sponsor: Kular Hospital (Other)
Responsible Party: Principal Investigator, Dr. Robert Rutledge, Research Director, Kular Hospital
Other Study IDs: TaBLFood-MGB
Record Dates: First submitted 2020-06-18; First posted 2020-06-22 (Actual); Last update posted 2020-06-22 (Actual); Status verified 2020-06

CONDITIONS: Obesity; Morbid Obesity; Bariatric Surgery Candidate; Food Selection; Diet Habit
MeSH Terms: conditions — Obesity; Obesity, Morbid; Food Preferences; Feeding Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mini-Gastric Bypass: Patients reported completing survey following Mini-Gastric Bypass
  Interventions: Other: Mini-Gastric Bypass

INTERVENTIONS:
Other: Mini-Gastric Bypass — Mini-Gastric Bypass bariatric surgery

SUMMARY:
Bariatric surgery (BS) has a history of new procedures and techniques arising and then disappearing due to problems and complications. The present is no different with new and old procedures changing with the regularity of night following day.

One of the important questions today in BS is the length and or need/value of the Biliopancreatic limb bypass (BPLL.) The Sleeve and the Band have "0" bypass, the RNY has a "short" bypass and the Biliopancreatic Diversion type procedures have a "long" (distal) bypass.

The Mini-Gastric Bypass Original Technique (MGB-OT) version of the One Anastomosis Bypass (OAGB) includes a "medium" length of bypass, longer than the BPLL of the RNY and shorter than the the "Long" BPL of the BPD procedures. In addition, uniquely, the MGB-OT includes a "Tailored" BPLL.

Not all OAGB surgeons use this approach and several have argued in favor of a "Fixed" BPLL of 150 cm.

This paper is part of a series of studies of the "Tailored" BPLL specifically in MGB-OT patients.

Notably it demonstrates in an online survey that patient reported weight loss and food choices change after MGB-OT and in addition the changes are related to the "Tailored" BPLL

DETAILED DESCRIPTION:
Introduction:

Studies of different Bariatric procedures have resulted in conflicting findings on the effects of the surgery on daily Dietary Food Choices (DFCs.) Some suggest a pure volume effect, others report changes in type and preferences and still others suggest the effects change over time. The Biliopancreatic Limb Length (BPLL) in the One Anastomosis Gastric Bypass (OAGB), Mini-Gastric Bypass-Original Technique (MGB-OT) version, includes a "tailored" BPLL. The purpose of this study was to investigate the relationship between BPLL and DFCs in patients undergoing MGB-OT. The primary hypothesis was that the changes in dietary habits and food choices would be related to the BPLL in the MGB-OT.

Methods:

Data from a long term online patient survey including MGB-OT patients were collected including basic demographics, MGB-OT BPLL, patient reported DFCs and weight loss classes. Linear regression modeling was used to assess the relative association between BPLL with various mean patient reported DFCs and a composite model of Food Choices.

Results:

Patients survey responses to be evaluated. Patients with reported BPLLs of 3 to 9 ft (92-274cm) will be selected. Patient reported mean weight loss classes to be evaluated. The linear relation to BPLL to be evaluated. The mean "Bad" Food Choices (BFC) to be determined.

Conclusions:

The present study of mean patient reported DFC outcomes following a "Tailored" BPLL in the MGB-OT version of the OAGB to be evaluated. The patient dietary food choices for fried foods, sugar sweetened beverages, processed meats and junk foods all to be determined. These changes linear regression to the Bilio-pancreatic limb length to be determined. In cases of the MGB-OT a longer Bilio-pancreatic Limb Length association with greater weight loss and a greater improvement in daily Dietary Food Choices would be major importance. The possibility of tailoring the power of a bariatric operation based upon BPLL might well be an important advancement in bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

* Post Mini-Gastric Bypass Patients

Exclusion Criteria:

-

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients completing survey following surgery for Mini-Gastric Bypass performed for morbid obesity
Sampling Method: Non-Probability Sample
Enrollment: 190 (Actual)
Dates: Start 2008-01-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Food Choices | from 1 year up to 10 years post operative Mini-Gastric Bypass
  Patient Reported Food choices

OTHER OUTCOMES:
Weight Loss | from 1 year up to 10 years post operative Mini-Gastric Bypass
  Pre and post reported weights and amount of reported weight loss

CONTACTS AND LOCATIONS:
Overall Officials: R Rutledge, MD, Principal Investigator — Kular Hospital
Locations (1):
- Kular Hospital, Khanna, Punjab, India

IPD SHARING:
Plan to Share IPD: No